CLINICAL TRIAL: NCT00127699
Title: Triple Dye Plus Alcohol Versus Triple Dye Alone for Newborn Umbilical Cord Care
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21353EP
Record Dates: First submitted 2005-08-05; First posted 2005-08-08 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Umbilical Cord; Infection
Keywords: Umbilical cord; Triple dye; Infant care
MeSH Terms: conditions — Infections | interventions — Ethanol

INTERVENTIONS:
Procedure: Alcohol swab of umbilical cord

SUMMARY:
In the United States (U.S.) there currently is no standard method of umbilical cord care, resulting in varying practices within and across institutions. These differences may result in an increase in morbidities for newborns such as the formation of umbilical granulomas and increases in acute care utilization. This study will determine which of two common methods of caring for newborn umbilical cords is superior - triple dye, followed by the application of rubbing alcohol, or triple dye alone.

DETAILED DESCRIPTION:
Infection of the umbilical cord of the newborn is a serious condition that can even lead to infant death. It has been well documented that the sources of infection among infants in hospitals is cross-contamination from other infants; S aureus is carried from infant to infant by nursery caregivers. Current and accepted cord care practices include aseptic techniques in cutting the umbilical cord, applying antimicrobial agents, hand washing, dry cord care and rolling the diaper below the cord to enhance drying (Evens, et. al, 2004).

Many studies have been performed to identify the best cord care practice. Zupan, et. al (2004) performed a meta-analysis of 21 studies that investigated cord care. Between all 21 studies many antimicrobial agents were used, including alcohol, triple dye, silver sulfadiazine, zinc powder, chlorhexidine, and salicylic sugar powder, along with dry cord care. It was identified that limited research has not shown a significant difference in outcomes between antimicrobial agent use and simply keeping the cord clean and dry. In high-income countries where mortality is low, important outcomes must include infections in the first month of life, maternal satisfaction, and time to cord separation. At the current time, there is no research that identifies the usefulness of applying colostrum, which has bacteriostatic properties, to the umbilical cord.

A prospective controlled trial was conducted by Golombek, S., et. al (2002) to compare only cord separation times between infants treated with triple dye as compared to alcohol. Of the 634 patients enrolled, one infant in the triple dye group was diagnosed with omphalitis; and one infant in the alcohol group was diagnosed with an ear infection. There was a statistically significant difference in cord separation time, with the alcohol group having a shorter separation time by 3 days (alcohol group 10 days, versus triple dye group 13 days) (p<0.0001). Nursing staff reported more satisfaction with alcohol alone. Parents universally expressed relief with cord separation in both groups.

Janssen, P., et al (2003) compared cord bacterial colonization and morbidity among newborns whose cords were treated with triple dye and alcohol versus dry cord care. Seven hundred sixty six infants were enrolled and randomized to a triple dye and alcohol group or a dry cord care group. Study groups were similar in all respects. Significantly more mothers in the dry care group stated that their infant's physician had mentioned concerns about infection to them compared with none in the triple dye group. There were no differences in reported rates of mothers contacting physicians in regard to concerns about infection. The most significant difference of observations of community health nurses between the two groups was periumbilical area exudates (p< 0.001) and foul odor (p<0.04) was more noticed in the dry cord care group. Though only one infant in the entire study developed omphalitis, which was in the dry cord care group, infants in the dry care group were significantly more likely to be colonized by E. coli, coag-neg staph, S. aures, and group B strep. Topical antimicrobial cord care may reduce bacterial colonization of the cord; there is no firm relationship between colonization and infection. Parents have expressed apprehension about cleaning the cord because of it's black appearance and brittle, rigid texture suggest that it will break off or hurt the infant if touched. Though not reported in scientific literature, increasing rates of breastfeeding may offer some protection to the newborn from infection. The study suggests that omphalitis remains a clinical entity and that there is potential risk in discontinuing bacteriocidal treatment of the umbilical cord stump. Cessation of bactericidal care of the umbilical stump must be accompanied by vigilant attention and education of parents to the signs and symptoms of omphalitis.

ELIGIBILITY:
Inclusion Criteria:

* Newborn admitted to the well-baby nursery
* >= 37 weeks gestation
* Born at Hershey Medical Center
* University Pediatric Associates patient

Exclusion Criteria:

* Baby with sepsis or admitted to the Neonatal Intensive Care Unit (NICU)
* <37 weeks gestation
* Not being followed by University Pediatric Associates

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2005-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Determine which of two common methods of caring for newborn umbilical cords is superior, triple dye followed by application of rubbing alcohol or triple dye alone

CONTACTS AND LOCATIONS:
Overall Officials: Alawia Suliman, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Result] Golombek SG, Brill PE, Salice AL. Randomized trial of alcohol versus triple dye for umbilical cord care. Clin Pediatr (Phila). 2002 Jul-Aug;41(6):419-23. doi: 10.1177/000992280204100607. PMID 12166794
- [Result] Janssen PA, Selwood BL, Dobson SR, Peacock D, Thiessen PN. To dye or not to dye: a randomized, clinical trial of a triple dye/alcohol regime versus dry cord care. Pediatrics. 2003 Jan;111(1):15-20. doi: 10.1542/peds.111.1.15. PMID 12509548
- [Result] Pezzati M, Biagioli EC, Martelli E, Gambi B, Biagiotti R, Rubaltelli FF. Umbilical cord care: the effect of eight different cord-care regimens on cord separation time and other outcomes. Biol Neonate. 2002 Jan;81(1):38-44. doi: 10.1159/000047182. PMID 11803175
- See also: Pediatric Clinical Research Office: Penn State Milton S. Hershey Medical Center — http://www.hmc.psu.edu/pedsclinicalresearch/index.htm